CLINICAL TRIAL: NCT06585228
Title: Detecting Cardiac Thrombi in Acute Ischemic Stroke on Cardiac CT Versus Transoesophageal Echocardiography (MtH-DETECT)
Brief Title: Detecting Cardiac Thrombi in Acute Ischemic Stroke on Cardiac CT Versus Transoesophageal Echocardiography
Acronym: MtH-DETECT
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jonathan Coutinho, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL84141.018.23
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke; Cardioembolic Stroke; Thrombus; Embolism; Left Atrial Thrombosis; Left Atrial Appendage Thrombosis
Keywords: Cardiac CT; Transoesophageal echocardiography; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Embolic Stroke; Thromboembolism | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Cardiac Computed Tomography — Cardiac CT acquired during the acute stroke imaging protocol
  Other Names: Cardiac CT; CCT
Diagnostic Test: Transesophageal echocardiography — Ultrasound through the oesophagus to assess cardiac structures.
  Other Names: TEE
Diagnostic Test: Repeated Cardiac Computed Tomography — A second cardiac CT performed after the TEE.
  Other Names: Cardiac CT

SUMMARY:
Rationale:

Cardiac CT acquired during the acute stroke imaging protocol (acute cardiac CT) has recently been shown to have a superior diagnostic yield than transthoracic echocardiography, which is currently the most commonly used method to screen for structural sources of cardioembolism in patients with acute ischemic stroke. The most common finding on acute cardiac CT are cardiac thrombi located in the left atrium (LA) and specifically the left atrial appendage (LAA). The higher diagnostic yield of acute cardiac CT compared to TTE is partially explained because CT allows for better visualization of the LAA, but also because cardiac thrombi may dissolve in the first days after stroke. Whether acute cardiac CT is the optimal diagnostic modality for LA thrombi in stroke patients is unknown, since data comparing it to transoesophageal echocardiography (TEE), which is the reference standard to detect LA thrombi, are lacking. The general hypothesis of this study is that acute cardiac CT is the optimal method to detect LA thrombi in ischemic stroke patients, since TEE can miss LA thrombi that dissolve in the first days after stroke.

Objectives:

1. Determine whether acute cardiac CT has a higher diagnostic probability of detecting LA thrombi compared to TEE or repeated cardiac CT in the subacute phase of ischemic stroke by assessing the rate at which LA thrombi dissolve in the first days after ischemic stroke occurrence.
2. Determine the positive predictive value of acute cardiac CT compared to TEE for the detection of LA thrombi. Study design: Prospective, single-centre, observational cohort Study population: 39 patients of 18 years or older with acute ischemic stroke and a LA thrombus detected on cardiac CT acquired during the acute stroke imaging.

Main study parameters/endpoints:

1. Rate at which LA thrombi visualized on acute cardiac CT dissolve in the first days after ischemic stroke.
2. False-positive rate for detection of left atrial thrombi on acute cardiac CT compared to TEE. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Clinical and imaging patient data which are obtained as part of standard care will be prospectively collected after written informed consent. Patient with a LA thrombus on acute cardiac CT will undergo TEE for research purposes after obtaining written informed consent. TEE is semi-invasive and associated with a small risk of major complications (<0.2%). Patients will also be exposed to additional radiation (1.4 mSV) due to sequential cardiac CT after TEE. The Radiation Dose Committee deemed this to be an intermediate risk. In a small minority of patients (<10%), another cardiac CT will be acquired 2 minutes after this sequential cardiac CT to ensure a clear, final assessment of the presence of an atrial appendage thrombus. This will result in a total additional radiation of 3 mSV for the two additional cardiac CT's. The Radiation Dose Committee deemed this to be an intermediate risk. As part of standard care, patients will be contacted for follow-up evaluation by a trained stroke nurse at 90 days. As a result of ischemic stroke, some patients become incapacitated to an extent they are unable to give informed consent. In these cases, the legal representative will be asked for informed consent. Decreased leveI of consciousness or aphasia are typical clinical characteristics of cardioembolic stroke. Therefore, it is pivotal to also include incapacitated acute ischemic stroke patients. Excluding these patients from the study would render the study non-representative of the study's target population (acute ischemic stroke patients with cardioembolic stroke due to LA thrombus).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of acute ischemic stroke
* Written informed consent from patient or representative
* Radiological diagnosis of cardiac thrombus in the LA, including the LAA, on cardiac CT acquired during the initial stroke imaging protocol.

Exclusion Criteria:

* Patients with a diagnosis other than acute ischemic stroke, such as: transient ischemic attack, intracerebral haemorrhage, subarachnoid haemorrhage, epilepsy, tumor.
* Absolute contraindication for TEE:

  * Perforated viscus
  * Esophageal stricture
  * Esophageal tumor
  * Esophageal perforation, laceration
  * Esophageal diverticulum
  * Active upper GI bleed
* Absolute contraindication for repeat cardiac CT

  * Documented previous severe reaction to iodinated contrast media, including anaphylaxis, angioedema and bronchospasm.
  * Severely impaired kidney function defined as estimated glomerular filtration rate of 30 mL/min/1.73 m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with acute ischemic stroke and a LA thrombus detected on cardiac CT acquired during the initial stroke imaging protocol at Amsterdam UMC, location AMC.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a left atrial thrombus | The assessment of a left atrial thrombus is performed when the patient arrives at the Emergency Department and undergoes the acute stroke imaging protocol including a cardiac CT.
  The proportion of patients with a LA thrombus detected on acute cardiac CT that dissolves in the first days after stroke, defined as thrombi that are seen on initial cardiac CT but are no longer visible on TEE and repeated cardiac CT.
Positive predictive value of acute cardiac CT compared to TEE. | The assessment of a left atrial thrombus is performed when the patient arrives at the Emergency Department and undergoes the acute stroke imaging protocol including a cardiac CT. The TEE is performed <7 days after the cardiac CT.
  Positive predictive value of acute cardiac CT compared to TEE.

SECONDARY OUTCOMES:
Other pre-defined high-risk and non-high-risk sources of embolism on cardiac CT and TEE | Cardiac CT is performed and assessed when the patients arrives at the Emergency Department. The TEE is performed <7 days after the cardiac CT.
  Other high-risk and non-high-risk sources that have been detected on cardiac CT and TEE.
Clinical impact of cardiac thrombi | The clinical data of patients with a thrombi is collected on arrival at the Emergency Department and follow-up is performed at 90 days and 2 years to assess functional outcome, recurrent stroke and cardiovascular events
  The clinical impact of detecting cardiac thrombi and other sources of embolism on acute cardiac CT and TEE, including any impact on stroke etiology according to Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Coutinho, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam University Medical Center (UMC), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided